CLINICAL TRIAL: NCT03884296
Title: Response to Live Attenuated Influenza Vaccine in Tonsillar Tissues and Blood
Acronym: FLU-Tonsil
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Not feasible to enroll participants
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Philip Grant, Assistant Professor of Medicine (Infectious Diseases), Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 50122; 5U19AI057229-15 (NIH)
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Influenza
Keywords: Obstructive sleep apnea; Quadrivalent live, attenuated influenza vaccine; Flumist
MeSH Terms: conditions — Influenza, Human; Sleep Apnea, Obstructive | interventions — FluMist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Study Phase (Other): Participants will be given the current year's quadrivalent, live, attenuated seasonal influenza vaccine (LAIV4)/FluMist® intranasally 3-14 days prior to tonsillectomy.
  Interventions: Biological: FluMist

INTERVENTIONS:
Biological: FluMist — Quadrivalent, live, attenuated influenza vaccine, intranasal spray

SUMMARY:
This is one project of a larger ongoing study related to the immune system's response to the flu virus. This study is designed to investigate the immune response to a nasal flu immunization in tonsillar tissue compared to what can be measured in the blood.

DETAILED DESCRIPTION:
This is a Phase IV study of licensed influenza vaccines with up to 50 male and female volunteers, 2-49 years of age. Volunteers were patients undergoing tonsillectomy for treatment of obstructive sleep apnea (OSA) or other non-infectious indication as part of their routine medical care.

The investigator intends to collect blood and lymphoid tissues routinely discarded during surgery from adults and children after routine seasonal live attenuated influenza vaccination (LAIV) to determine how immune memory develops at the actual site of infection, and how immunization may alter this process.

The first research study visit will take place approximately 3-14 days prior to the scheduled date of tonsillectomy surgery. During this visit, 20 mL blood sample will be obtained and participants will receive FluMist (intranasal, quadrivalent, live-attenuated influenza vaccine). This is one of the routinely available and recommended vaccines for the age groups included in this study.

The second study visit will take place on the same day of the scheduled surgery for the tonsillectomy. Another blood sample (maximum volume of 20 mL) will be collected along with the discarded tonsillar tissue. Blood and tissues will be sent to the lab.

ELIGIBILITY:
Inclusion Criteria:

1. 2-49-year-old male and female patients undergoing tonsillectomy for obstructive sleep apnea or other non-infectious indication.
2. Willing and able to complete the informed consent process
3. Availability for follow-up for the planned duration of the study
4. Acceptable medical history by review of inclusion/exclusion criteria

Exclusion Criteria:

1. Prior off-study vaccination with seasonal influenza vaccine within three months of study vaccination
2. Life-threatening reactions to previous influenza vaccinations
3. Asthma (contraindication for receipt of LAIV4)
4. Allergy to egg or egg products or to vaccine components including gentamicin, gelatin, arginine or MSG.
5. Active systemic or serious concurrent illness, including febrile illness on the day of vaccination
6. History of immunodeficiency (including HIV infection)
7. Known or suspected impairment of immunologic function; may include significant liver disease, diabetes mellitus treated with insulin or moderate to severe renal disease
8. Hospitalization in the past year for congestive heart failure or emphysema.
9. Chronic Hepatitis B or C.
10. Recent or current use of immunosuppressive medication, including systemic glucocorticoids (corticosteroid nasal sprays and topical steroids are permissible). Use of oral steroids (<20mg prednisone-equivalent/day) may be acceptable after review by the investigator.
11. Participants in close contact with anyone who has a severely weakened immune system
12. Malignancy, other than squamous cell or basal cell skin cancer (includes solid tumors such as breast cancer or prostate cancer with recurrence in the past year, and any hematologic cancer such as leukemia).
13. Autoimmune disease (including rheumatoid arthritis treated with immunosuppressive medication such as Plaquenil, methotrexate, prednisone, Enbrel) which, in the opinion of the investigator might jeopardize volunteer safety or compliance with the protocol.
14. History of blood dyscrasias, renal disease, or hemoglobinopathies requiring regular medical follow up or hospitalization during the preceding year
15. Use of any anti-coagulation medication such as Coumadin or Lovenox, or anti-platelet agents such as aspirin (except up to 325 mg. per day), Plavix, or Aggrenox will be reviewed by investigators to determine if study participation would affect the volunteer's safety or compliance with the protocol.
16. Receipt of blood or blood products within the past 6 months or planned used during the study.
17. A medical or psychiatric condition or occupational responsibilities that preclude participant compliance with the protocol
18. Receipt of an inactivated vaccine 14 days prior to study enrollment, or planned vaccinations prior to completion of last study visit (~ 14 days after study vaccination)
19. Receipt of a live, attenuated vaccine within 60 days prior to enrollment of planned vaccination prior to completion of last study visit (~ 14 days after study enrollment)
20. Need for allergy immunization (that cannot be postponed) until after the last study visit.
21. History of Guillain-Barre# syndrome
22. Pregnant or breastfeeding woman
23. Use of investigational agents within 30 days prior to enrollment or planned use during the study.
24. Donation of the equivalent of a unit of blood within 6 weeks prior to enrollment or donation of platelets within 2 weeks of enrollment or planned donation prior to completion of the last visit.
25. Any condition which, in the opinion of the investigator, might interfere with volunteer safety, study objectives or the ability of the participant to understand or comply with the study protocol.

Ages: 2 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Plasma HAI titer | Day 3-14 after receipt of LAIV
  HAI titer measures imune response to influenza vaccination
Number of Participants With Related Adverse Events | Day 0 to 14 post-immunization
  We will capture AEs to LAIV

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University Medical Center, Lane building L134, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No